CLINICAL TRIAL: NCT06252467
Title: Effects of Photobiomodulation Therapy on Performance in Successive Time-to-Exhaustion Cycling Tests: A Randomized Double-Blinded Placebo Controlled Trial
Brief Title: Photobiomodulation Therapy on Performance in Successive Cycling Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Aurélio Vaz, PhD (Other)
Responsible Party: Sponsor-Investigator, Marco Aurélio Vaz, PhD, Head of Neuromuscular Plasticity Laboratory and Principal Investigator, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 708.362
Record Dates: First submitted 2023-11-14; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Photobiomodulation Therapy; Cyclists; Performance
Keywords: Phototherapy; VO2 response; muscle oxygenation; cyclists; performance
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
  Crossover, randomized, double-blind trial (blinding of the cyclists and the researcher responsible for evaluations)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Device: Active Photobiomodulation Therapy Phototherapy treatment (Photobiomodulation therapy or placebo) was performed using a Photobiomodulation therapy device (Vectra Genisys Systems, Chattanooga Group, Dallas, TX, USA). The cluster probe consisted of five low-level laser therapy diodes (850 nm) and 28 light emitting diodes therapy (670 nm, 880 nm, and 950 nm). Photobiomodulation therapy was applied in nine sites of each quadriceps femoris muscle
  . A dosage of 15 J per site led to a total energy of 135 J per thigh, effectively increasing cycling performance in a previous study. We chose to apply Photobiomodulation therapy specifically to the quadriceps femoris because this muscle group is of utmost significance in generating torque and propelling the pedaling cycle. Its pivotal role in cycling performance made this muscle a prime target for the Photobiomodulation therapy intervention in our study.
  Interventions: Device: Photobiomodulation Therapy
- Placebo Comparator (Placebo Comparator): Device: Placebo Photobiomodulation The placebo treatment was performed in exactly the same manner as the Photobiomodulation therapy treatment, but with the device switched off, and the cluster was held stationary in contact with the skin at a 90° angle, with light pressure on the skin. The total application time of Photobiomodulation therapy or placebo was ~5 min for both limbs (9 points per thigh = 18 points × 16 s per point) before each time-to-exhaustion test.
  Interventions: Device: Placebo Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation Therapy — Phototherapy treatment (Photobiomodulation therapy or placebo) was performed using a Photobiomodulation therapy device (Vectra Genisys Systems, Chattanooga Group, Dallas, TX, USA). The cluster probe consisted of five low-level laser therapy diodes (850 nm) and 28 light emitting diodes therapy (670 nm, 880 nm, and 950 nm). Photobiomodulation therapy was applied in nine sites of each quadriceps femoris muscle
  . A dosage of 15 J per site led to a total energy of 135 J per thigh, effectively increasing cycling performance in a previous study. We chose to apply Photobiomodulation therapy specifically to the quadriceps femoris because this muscle group is of utmost significance in generating torque and propelling the pedaling cycle. Its pivotal role in cycling performance made this muscle a prime target for the Photobiomodulation therapy intervention in our study.
  Arms: Active Comparator
Device: Placebo Photobiomodulation — The placebo treatment was performed in exactly the same manner as the Photobiomodulation therapy treatment, but with the device switched off, and the cluster was held stationary in contact with the skin at a 90° angle, with light pressure on the skin. The total application time of Photobiomodulation therapy or placebo was ~5 min for both limbs (9 points per thigh = 18 points × 16 s per point) before each time-to-exhaustion test.
  Arms: Placebo Comparator

SUMMARY:
The goal of this study was to investigate the effects of Photobiomodulation therapy (PBMT) on performance, oxygen uptake (VO2 kinetics), and lower limb muscle oxygenation during three successive time-to-exhaustion tests (TTEs) in cyclists. This was a double blind, randomized, crossover, placebo-controlled trial study. Sixteen cyclists (~23 years old), with a cycling training volume of ~460 km/week, volunteered for this study. In the first session, cyclists performed a maximal incremental test to determine maximal oxygen uptake and maximal power output (POMAX). In the following sessions, cyclists performed three consecutive TTEs at POMAX. Before each test, PBMT (135 J/thigh) or a placebo (PLA) PBMT was applied to both thighs. VO2 amplitude, O2 deficit, time delay, oxyhemoglobin (O2Hb), deoxyhemoglobin (HHb), and total hemoglobin (tHb) were measured during tests on the right vastus lateralis. The PBMT, applied before three successive TTE, increased performance of the first and second TTE (~10-12%) tests, speed of VO2 and HHb kinetics during the first test, and increased peripheral muscle oxygenation (increase in HHb and tHb) in the first and second exhaustion tests. However, the PBMT effects were attenuated in the third TTE, as performance and all the other outcomes were similar to the ones from the PLA intervention. In summary, PBMT application increased the first and second successive TTEs, speed of VO2, and muscle oxygenation.

DETAILED DESCRIPTION:
The goal of this study was to investigate the effects of Photobiomodulation therapy (PBMT) on performance, oxygen uptake (VO2 kinetics), and lower limb muscle oxygenation during three successive time-to-exhaustion tests (TTEs) in cyclists. Our study was characterized as a crossover, randomized, double-blind trial (blinding of the cyclists and the researcher responsible for evaluations). All protocols were explained to the participants, who voluntarily provided their consent to participate in the investigation through an informed consent document. This study received approval from the Research Ethics Committee for Human Subjects Studies at the institution where the research was conducted (number 708.362). Inclusion criteria involved cyclists aged 18-30 years, with a competitive history and no history of musculoskeletal injuries in the lower limbs in the last two years. Exclusion criteria included chronic disease, smoking, metabolic disorders, use of steroids in the last six months, chronic disease, physical disabilities, and use of antibiotic drugs in the previous week. The cyclists participating in the present study had ~6.5 years of regular training/competition and no history of lower limb muscular and/or skeletal injuries. Each cyclist visited the laboratory on three occasions. At the first visit, cyclists performed a maximum incremental test and familiarization to three successive TTEs. At the two subsequent visits, participants performed a standard protocol of three successive TTEs at maximal power output (POMAX) with preferred cadence, and PBMT or placebo (PLA) treatments were applied before each trial. The three testing days were performed with a 72h interval apart. A single therapist was involved with the random allocation of the PBMT and PLA interventions. This therapist received instructions not to disclose the treatment modality employed during each assessment session to either the cyclists or other researchers involved with data collection and data analysis. Furthermore, cyclists utilized opaque eyewear to shield their eyes and obstruct their visual access (visual blinding) during the PBMT or PLA intervention. The therapist was explicitly advised against revealing the treatment modality to both the cyclists and the other researchers. PBMT did not elicit any thermal or tactile sensations, thereby ensuring that athletes remained unaware of the specific application on their thigh area. The random assignment was determined through a basic drawing of lots during the first testing session, determining the allocation of either active PBMT or inactive PLA.

ELIGIBILITY:
Inclusion Criteria:

* Cyclists aged 18-30 years;
* Competitive history;
* No history of musculoskeletal injuries in the lower limbs in the last two years.

Exclusion Criteria:

* Chronic disease;
* Smoking;
* Metabolic disorders;
* Use of steroids in the last six months;
* Physical disabilities;
* Use of antibiotic drugs in the previous week.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Cycling performance | Cyclits performed a standard protocol of three successive tests to exhaustion at maximal power output with preferred cadence, and photobiomodulation therapy or placebo treatments were applied before each trial. The three testing days were performed
  Cyclists performed the three successive time-to-exhaustion at maximal power output at their preferred cadence. Exhaustion was defined as the time when the cyclist was unable to maintain a cadence above 70 rotations per minute. During the successive time-to-exhaustion, cadence and power output were measured using the cycle ergometer software (Excalibur Sport, Lode Medical Technology, Groningen, Groninga, The Netherlands). The cyclists' evaluation was conducted utilizing a cycle ergometer (Excalibur Sport, Lode Medical Technology, Groningen, Groninga, The Netherlands) configured to match their bike's handlebar and seat settings.
Oxygen uptake | Oxygen uptake response was measured during the three sucessive time-to-exhaustion in two days (Photobiomodulation Therapy or Placebo) with a 72 hours interval apart.
  Oxygen uptake was measured breath-by-breath using an open-circuit gas analyzer (Quark CPET, Cosmed, Rome, Lazio, Italy). Oxygen uptake measurements were plotted to facilitate the exclusion of values lying beyond four standard deviations above or below the average of the dynamic window (three breaths), taken as the reference for the overall curve average. Analysis of oxygen uptake kinetics during successive time-to-exhaustion was converted into 5 seconds windows, and mean values were calculated. The analysis of oxygen uptake kinetics was dependent on the duration of the three time-to-exhaustion for each athlete in each condition (Photobiomodulation therapy or placebo). Oxygen uptake kinetics were calculated with the nonlinear least-squares method implemented in MATLAB (Mathworks, Natick, MA, USA) to adjust the oxygen uptake data.

SECONDARY OUTCOMES:
Periphery muscle oxygenation | Periphery muscle oxygenation response was measured during the three sucessive time-to-exhaustion in two days (Photobiomodulation Therapy or Placebo) with a 72 hours interval apart.
  Peripheral muscle oxygenation data collection was performed using a NIRS (PortaMon, Artinis Medical Systems, Elst, Guéldria, Netherlands) probe (light emitting and photoreceptor), which was positioned in the vastus lateralis muscle belly of the right lower limb, longitudinally located between the femur's lateral epicondyle and trochanter, fixed with adhesive tape (3M Company, Saint Paul, MN, USA), and wrapped by the cyclist's bretelle to prevent light penetration during all time-to-exhaustion. Data from the NIRS system were analyzed from average windows every 20% of the time-to-exhaustion tests and retests. The oxyhemoglobin, deoxyhemoglobin, and total hemoglobin were evaluated. Furthermore, oxyhemoglobin, deoxyhemoglobin, and total hemoglobin values were normalized by their respective mean values obtained at rest before the first time-to-exhaustion in each condition, which were used to compare the experimental situations (Phobiomodulation Therapy or Placebo).

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Aurélio Vaz, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No